# Statistical Analysis Plan: GCA-SAP-2019-001-01 for T-PLUS Trial

Ascensia Diabetes Care Global Clinical Affairs

Reference Protocol:

Protocol Title:

GCA-PRO-2019-001-01

User Performance of the T-PLUS Blood Glucose Monitoring Systems



The statistical plan is intended to satisfy requirements for clinical study data analyses in:

FDA (2018) Self-Monitoring Blood Glucose Test Systems for Over-the-Counter Use, Draft Guidance for Industry and Food and Drug Administration Staff, Issued 30Nov2018,

ISO 15197:2013 In vitro diagnostic test systems – Requirements for blood-glucose monitoring systems for self-testing in managing diabetes mellitus, 2<sup>nd</sup> Ed. 2023-05-15 (section 8)

# **ABBREVIATIONS**

| Abbreviation | Interpretation |
|------------------------|--------------------------------------|
| Adj. R <sup>2</sup> | Adjusted R Squared |
| BG | Blood Glucose |
| CAP | Capillary |
| Cum. | Cumulative |
| DM | Diabetes Management |
| Eval | Evaluable |
| GCA | Global Clinical Affairs |
| GE | Greater Than or Equal To |
| HbA1c | Hemoglobin A1c |
| HCT | Hematocrit |
| ISO | International Standards Organization |
| LCL | Lower Confidence Limit |
| LL | Lower Limit |
| Lower CI | Lower Confidence Limit |
| LT | Less Than |
| Max | Maximum |
| Min | Minimum |
| N | Sample Size |
| NA | Not Applicable or No Answer |
| PRO | Protocol |
| PWD | Person with Diabetes |
| RH | Relative Humidity |
| SD, Std Dev | Standard Deviation |
| SE, Std Err, Std Error | |
| STAFF | Site Staff |
| SUB | Subject |
| Sy.x | Root Mean Square Error |
| Temp | Temperature |

## 1. Sample Size

1.1 ISO 15197:2013 Objective – Accuracy in People with Diabetes

Let MeterBG = meter blood glucose result;

LabBG = laboratory method (YSI) comparator blood glucose result.

D = MeterBG - LabBG

RD = 100\*(MeterBG - LabBG) / LabBG

Assume 315 evaluable results from people with diabetes. The ISO 15197:2013 acceptance criterion is that 95% of those evaluable results must satisfy the accuracy criteria:

 $|D| = |MeterBG - LabBG| \le 15 \text{ mg/dL}, \text{ for LabBG} < 100 \text{ mg/dL}$  or

 $|RD| = 100*|MeterBG - LabBG| / LabBG \le 15\%$ , for LabBG  $\ge 100 \text{ mg/dL}$ .

With n = 315, Xc = 300 results would be required to satisfy the accuracy criteria. At  $P_0 = 96.79\%$ , there is approximately a 95% chance of satisfying the ISO objective. Conversely, at  $P_a = 92.77\%$ , there is approximately a 95% chance of failing to satisfy the ISO objective.

1.2 FDA Objective – Accuracy with All Subjects Included

For the FDA accuracy objective, a result (MeterBG) is considered accurate if:

 $|RD| = 100*|MeterBG - LabBG| / LabBG \le 15\%$ , regardless of the value of LabBG.

Assuming n = 350 evaluable results, Xc = 333 results would be required to satisfy the accuracy criteria. At  $P_0 = 96.65\%$ , there is approximately a 95% chance of satisfying the FDA 15% objective. Conversely, at  $P_a = 92.81\%$ , there is approximately a 95% chance of failing to satisfy the FDA accuracy objective.

The FDA guidance has a second criterion, that 99% of n evaluable results must have  $|RD| \le 20\%$ . Inasmuch as the two criteria are considered separately, there is no consideration for multiplicity. For the n = 350, the 20% criterion requires a critical value of Xc = .99\*350

= 346.5  $\rightarrow$  347. For this critical value and sample size, with P<sub>0</sub> = 99.61%, there is approximately a 95% chance of satisfying the FDA 20% criterion. Conversely, there is approximately a 95% chance of failing to satisfy the 20% criterion if the chance of obtaining a result within  $\pm 20\%$  of corresponding comparator measurement is only 97.8%.

Note that each glucose result obtained with the evaluation device will be considered either 'accurate' or 'not accurate', where accuracy depends on the particular test criterion.

## 1.3 Internal Objective

For subjects with diabetes only (PWDs):

The criterion is defined to be:

 $|D| \le 12.5 \text{ mg/dL if LabBG} < 100 \text{mg/dL, or:}$ 

 $|RD| \le 12.5\%$  if LabBG  $\ge 100$ mg/dL

The hypothesis:

 $H_0$ : Pr{criterion met} < 95%

will be tested against the alternative:

 $H_1$ : Pr{criterion met}  $\geq 95\%$ 

With n = 315, the critical value is Xc = 294 yields a power to reject H0 if Pr{criterion met} = 0.95 is ~92.63%.

Table 1.1 summarizes the power statements made in 1.1, 1.2, and 1.3.

| Table 1.1 1 twee Statements for 150 and 1 DA Acceptance Circuia | | | | | | | |
|---|---|---|---|---|---|---|---|
| Criterion | erion N Xc Po* Pr{PASS Po} Pa** Pr{FAIL Pa} | | | | | | |
| ISO | 315 | 300 | 96.79% | 95.02% | 92.77% | 94.95% | |
| ±12.5 | 315 | 294 | 95.00% | 92.63% | 90.60% 94.64% | | |
| FDA-15% | 350 | 333 | 96.65% | 95.00% | 92.81% | 94.95% | |
| FDA-20% | 350 | 347 | 99.61% | 95.05% | 97.80% | 95.00% | |
| *Po is the | mini | imun | n required | (hypothetical | ) probab | oility that any mea | surement |
| would me | et th | e de | finition of | an "accurate" | result, i | n order to have | |
| approxim | ately | a 95 | % chance t | hat at least Xo | out of N | l results would be | 9 |
| "accurate" (PASS) | | | | | | | |
| **Pa is the | **Pa is the maximum required (hypothetical) probability that any measurement | | | | | | |
| would meet the definition of an "accurate" result, in order to have | | | | | | | |

approximately a 95% chance that fewer than Xc out of N results would be

Table 1.1 Power Statements for ISO and FDA Acceptance Criteria

In general, critical values depend on actual sample size. The sample size and associated critical values for accuracy tests (the minimum required numbers of "accurate" results) are determined by regulatory guidance. The values of Po and Pa are affected by actual sample size.

## 2. Blood Glucose Measurements

"accurate" (FAIL)

Some data analysis follows analyses and presentations described in ISO Section 15197:2013, Section 8. See Table 3 for scheme of data analysis, including capillary blood and venous blood.

Other data analysis follows analyses and presentations described in the FDA 2018 OTC Guidance. See Table 4 for scheme of FDA 2018 OTC data analysis, including capillary blood and venous blood.

Blood glucose measurements will all be made in units of mg/dL. Graphs (other than error grids) involving blood glucose concentrations will be constructed in both mg/dL and mmol/L (for ISO analyses; analyses for FDA reporting will include tables and graphs in mg/dL only). The conversion of X mg/dL to Y mmol/L will be as follows:

$$Ymmol / L = \frac{Xmg/dL}{18.016}$$

Linear regression will be performed on data comparisons as shown in Tables 6.1 and 6.2.

**Modified Bland-Altman Plots** – Modified Bland-Altman plots (difference between evaluation device results and reference results plotted against reference results) will be constructed for all comparisons described in Tables 6.1 and 6.2.

#### 3. Accuracy Analyses

## 3.1 ISO Objective

At least 95% of the glucose results obtained using the evaluation device must be accurate, namely:

$$-15\% \le RD \le +15\%$$
  $LabBG \ge 100mg / dL$ 
OR

$$-15mg/dL \le D \le +15mg/dL$$
  $LabBG < 100mg/dL$ 

As discussed in section 0 (Sample Size), with n =315, the critical number (minimum) of accurate results is 300, which yields approximately a 95% chance of satisfying the ISO objective criterion if the actual probability that any result will be accurate is at least 96.79%. Symbolically, the ISO criterion is equivalent to testing the hypothesis:

$$H_0: \text{Prob}\{accurate\} < 96.79\%$$

versus the alternative:

$$H_1: \text{Prob}\{accurate\} \ge 96.79\%$$

There is approximately a 95% chance that the null will NOT be rejected if the actual probability that a result with the evaluation device would satisfy this definition of accuracy is only about 92.76%.

#### 3.2 Venous Goal

Venous glucose results will be analyzed in the same fashion as the ISO accuracy objective for subject-generated capillary (fingerstick) results for only evaluable results from subjects with diabetes, and the same acceptance criteria applied.

## 3.3 FDA Objectives

## 3.3.1 95% within ±15%

With n = 350, at least Xc = 333 measurements must be within  $\pm 15\%$  of LabBG. This requirement is equivalent to testing the hypothesis:

$$H_0$$
:  $\Pr\{|RD| \le 15\%\} < 0.9664$ 

against the hypothesis:

$$H_1$$
:  $\Pr\{|RD| \le 15\%\} \ge 0.9664$ 

with  $Pr\{reject H_0|p=0.9664\} \approx 0.9488$ 

## 3.3.2 99% within ±20%

With n = 350, at least Xc = 347 measurements must be within  $\pm 20\%$  of LabBG. This requirement is equivalent to testing the hypothesis:

$$H_0$$
:  $\Pr\{|RD| \le 20\%\} < 0.9960$ 

against the hypothesis:

$$H_1$$
:  $\Pr\{|RD| \le 20\%\} \ge 0.9960$ 

with  $Pr\{\text{reject } H_0 | p=0.9960\} \approx 0.9466$ 

## 3.4 Internal Accuracy Objective

The criterion is defined to be:

$$|D| \le 12.5 \text{ mg/dL if LabBG} < 100 \text{mg/dL, or:}$$

$$|RD| \le 12.5\%$$
 if LabBG  $\ge 100$ mg/dL

The hypothesis:

$$H_0$$
: Pr{criterion met} < 95%

will be tested against the alternative:

$$H_1$$
:  $Pr\{criterion\ met\} \ge 95\%$ 

With n = 350, the critical value is Xc = 327 yields a power to reject H0 if Pr{criterion met} = 0.95 is ~0.9246.

### 3.4.1 Study-Staff-Generated Capillary Testing Goal

Study-staff-generated capillary results will be analyzed in the same fashion as the ISO accuracy objective for subject-generated capillary (fingerstick) results for only evaluable results from subjects with diabetes, and the same acceptance criteria applied.

Study-staff-generated capillary results will be analyzed in the same fashion as the FDA accuracy objective for subject-generated capillary (fingerstick) results for only evaluable results from ALL subjects, and the same acceptance criteria applied.

## 3.5 Some Additional Comments about Hypothesis Tests

Power and risk calculations were made based on the assumption that n = 315 for the ISO accuracy objective, and for n = 350 for the FDA accuracy objective. It is possible that the total number of results may differ from the minimum requirement, depending on the numbers of subjects actually enrolled and the number of evaluable results. The critical value is always 95% of the total sample size of evaluable results. However, power statements made earlier were based on n = 315 or n = 350, so these statements may only be approximate.

No adjustment will be made for multiplicity. Each test will be evaluated without regard to the results of any other test.

## 3.6 By-Site Analyses

Only one site will be included in this study, so there will be no specific "by site" analyses.

3.7 Descriptive Statistics on Differences (D) and Relative Differences (RD) from Reference Descriptive statistics: mean (average), standard deviation, median, minimum, and maximum of D (LabBG < 100 mg/dL) and RD (LabBG ≥ 100 mg/dL), will be computed.

## 3.8 Confidence Intervals

Confidence intervals (95%, two-sided) for all ISO and FDA objective proportions (percents) will be computed using the Clopper-Pearson<sup>1</sup> (1934) formula:

$$P_L = \frac{X * F_{\alpha/2}^{-1}(2X, 2(n-X+1))}{n-X+1+X * F_{\alpha/2}^{-1}(2X, 2(n-X+1))}$$

-

<sup>&</sup>lt;sup>1</sup> Clopper, C.J., Pearson, E.S. (1934) The use of confidence or fiducial limits as illustrated in the case of the binomial, Biometrika, 26, 404-413

and:

$$P_U = \frac{X * F_{1-\alpha/2}^{-1}(2X, 2(n-X+1))}{n-X+1+X * F_{1-\alpha/2}^{-1}(2X, 2(n-X+1))}$$

 $P_L$  = lower limit

 $P_U = upper limit$ 

X = number of "accurate" results (per the relevant definition of "accurate")

## 3.9 Error Distributions

The numbers and percents of values of D (LabBG < 100 mg/dL) falling within  $\pm 5$ ,  $\pm 10$ ,  $\pm 15$ , and  $\pm 20$  mg/dL, and the numbers and percents of values of RD (LabBG  $\geq 100$  mg/dL) falling within  $\pm 5$ ,  $\pm 10$ ,  $\pm 15$ , and  $\pm 20$  percent will be tabulated.

## 4. Regression, Modified Bland-Altman Plots, Radar Plot, and Outlier Analysis

## 4.1 Weighted Least Squares (WLS)

A linear regression of the meter results (MeterBG) against the YSI reference method results (LabBG) via weighted least squares (WLS) will be performed, with weights:

$$w = \frac{1}{YSI^2}$$

used to account for the proportional variance nature of blood glucose measurements (Draper and Smith, 1998)<sup>2</sup>.

## 4.2 Studentized Residuals and Outlier Identification

Studentized residuals from the regression will be computed, i.e.,

<sup>2</sup> Draper, N. R., Smith, H., (1998) Applied Regression Analysis, 3rd Ed., John Wiley and Sons

$$e_i = y_i - \hat{y}_i$$

$$\varepsilon_i = \frac{e_i}{s_e \sqrt{1 - h_{ii}}}$$

That is, a studentized residual,  $\varepsilon$ , is the residual, e, divided by the standard error,  $s_e \sqrt{1 - h_{ii}}$ , of the residual. The variables  $h_{ii}$  are the diagonal elements of the "hat" matrix:

$$H = X[X'W^{-1}X]^{-1}X'W^{-1}$$

The matrix W is a diagonal matrix with the regression weights,  $w = \frac{1}{YSI^2}$  on the diagonal.

A meter result will be considered an "outlier" if its corresponding studentized residual is outside the interval  $(\Phi^{-1}(0.005), \Phi^{-1}(0.995)) \approx (-2.576, +2.576)$ , corresponding to a 99% interval for a standard normal variate. The function  $\Phi^{-1}(p)$  is the inverse cumulative distribution function of a standard normal random variable; that is, the function is a z-score.

Confidence bands (99%) for the regression (individual) predictions will be computed. Scatter plots of MeterBG vs. LabBG will be constructed, with the regression line, the confidence bands, and the line of identity (Y = X) will all be plotted.

#### 4.2 Modified Bland-Altman Plots

A Modified Bland-Altman Plot, with D plotted against LabBG (no limits on the range), will be constructed for subject-generated fingerstick, staff-generated fingerstick, and venous results. The limits for accuracy of individual results, per ISO:15197:2013, will also be plotted on the graphs.

#### 4.3 Radar Plots

Radar plots will be made. Two plots (one with units of mg/dL and one with units of mmol/L) will be constructed using only PWD data (ISO), and will include ISO 15197:2013 bifurcation of criteria (difference for YSI < 100 mg/dL, relative difference when YSI ≥ 100 mg/dL). Another plot will be constructed for all evaluable data (FDA) in mg/dL.

## 5. Error Grid Analyses

Parkes consensus error grids will be constructed for combined strip lots, and combined sites as described in Tables 6.1 and 6.2. There is no criterion for percentage of values within the error grid zones.

# 6. Data Analysis Schemes

Table 6.1 -Data Analysis Scheme (per ISO15197:2013)

| Blood<br>Type | Data<br>Comparison | Regression<br>Tables | Bland<br>Altman<br>Plots | Accuracy | Error<br>Grid | Error Interval tables (5,10,15, 20, >20%) |
|---|---|---|---|---|---|---|
| Capillary | Subject vs. YSI | <b>X</b> * | X*** | X* | <b>x</b> * | X* |
| | Staff vs YSI | <b>X</b> * | X*** | <b>X</b> * | <b>x</b> * | X* |
| Venous | Results vs. YSI | x* | X*** | x* | x* | x* |

<sup>\*</sup> Combined sites

Table 6.2 -Data Analysis Scheme (per draft FDA OTC Guidance 2018)

| Blood<br>Type | Data<br>Comparison | Regression<br>Tables | Scatter<br>Plots | Accuracy | Error<br>Grid | Error Interval tables (5%,7%,10%,15%,20%) |
|---|---|---|---|---|---|---|
| Capillary | Subject vs.<br>YSI | X* | X*** | X* | x* | x* |
| | Staff vs YSI | <b>X</b> * | X*** | X* | <b>X</b> * | x* |

<sup>\*</sup> Combined sites

Note – Samples outside +/- 20% will be identified and listed (per draft FDA 2018).

<sup>\*\*\*</sup> Plots with different symbols denoting whether observations are outliers

<sup>\*\*\*</sup> Plots with different symbols denoting whether observations are outliers

## 7. Subject Questionnaires

## 7.1 *Questionnaire 1 – Ease of Use*

Subject questionnaire 1 will consist in part of questions/statements for which a numerical score or rating (1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree) will be provided by the subjects and entered by the study staff. For these numerically-scored questions, frequency distributions will be tabulated. For PWD subjects only (ISO 15197:2013 requirements), hypothesis tests for selected statements will be performed. The hypotheses are:

 $H_0$ :  $Pr\{response \ge 3\} < 90\%$  versus the alternative:

$$H_a$$
:  $Pr\{response \ge 3\} \ge 90\%$ 

The critical number of responses greater than or equal to 3, Xc, is a function of the actual sample size, and will be chosen such that  $0.95 = \sup Pr\{X \ge X_c | 100p\% = 90\%\}$ . For example, if n = 315, then Xc = 276, so that  $Pr\{X \ge X_c | 100p\% = 90\%\} \approx 0.9299 \le 0.95$ . That is, 276 is the number of responses  $\ge 3$  which yields the largest value of  $Pr\{X \ge X_c | 100p\% = 90\%\} \le 0.95$  for n = 315.

## 7.2 Questionnaire 2, Diabetes Management

Frequencies of responses will be tabulated for statements/questions in the Diabetes Management Questionnaire.

## 8. Demographic, Diabetes History, Medications and Disease State Data

Descriptive statistics for subject Demographic, Diabetes History, Medications and Disease State data will be computed as appropriate. Histograms will be constructed where appropriate. A percentage of subjects < 65 years of age will be calculated.

#### 9. Other Tables

## 9.1 Hematocrit Analysis

Hematocrit will be measured in singlet for each subject. For ISO 15197 analyses, subjects with a hematocrit determination that is out of range (outside the range 0-70%) cannot be used for blood glucose measurement comparisons.

The mean, median, minimum, maximum, and standard deviation, will be computed for hematocrit determinations.

## 9.2 Temperature and Humidity

Mean, median, standard deviation, minimum and maximum room temperature and humidity will be computed.

#### 9.3 Glucose Distribution

The distribution of YSI glucose and a histogram (combined sites) for both capillary and venous blood will be provided. The mean, median, minimum, maximum, and standard deviation, will be computed for glucose distributions, by site and for both sites combined.

In addition, the number of capillary samples with concentrations <80 and > 250 mg/dL will be reported.

## 10. Data Listing

A listing of the data (excel sheet) is needed for the clinical study report. The listing should include: subject and staff fingerstick meter results, venous meter results, AST results, capillary and venous YSI results, subject ID, hematocrit.

## 11. Data Evaluability

Blood glucose data will be considered <u>not</u> evaluable for the following reasons:

- Subjects with either no hematocrit result or a hematocrit result outside of meter specifications (0-70%) (for FDA accuracy analyses, there is no requirement to have a hematocrit value; this requirement only pertains to ISO analyses).
- BG readings from **subject** meter tests that the <u>subject</u> feels were incorrectly completed. (If the subject states that the test s/he performed was completed incorrectly, and repeats the test, then the new BG reading will be used as the subject test.) Tests of each type (e.g., subject fingerstick) made be performed up to 3 times, i.e., repeated up to 2 times if the tester feels that the test was performed improperly.

- Failure to separate the plasma from the red cells (for YSI analysis) within 15 minutes of obtaining the corresponding evaluation meter result.
- Discrepant YSI replicate results will be excluded<sup>†</sup>. The comparator value for the subject will be the average of the non-outlier replicates. Should only a single replicate value be obtained for a given subject, it will be used as the comparator value.
- Subject plasma samples that do not have in-range serum controls tested after subject plasma test will be considered non evaluable.

Note: If supplemental or unplanned analyses are requested they will be presented in a supplemental report.

\_

<sup>†</sup> Glucose values of the YSI replicates should be within  $\pm 4$  mg/dL when average of replicates < 100 or  $\pm 4\%$  of each other when average of replicates  $\geq 100$ ; if not, an additional assay should be run.

## 12. Laboratory Instrument Quality Control

Runs using serum control material at multiple levels will be executed daily for each laboratory glucose comparator instrument used in the study. The run means will be compared to lower and upper limits for each level. If the minimum and maximum value of individual measurements are within lower and upper limits, the run means do not need to be compared to those limits also.

A regression line will be fit using the instrument results regressed against target values as set by Ascensia Diabetes Care analytical laboratory. For levels with target values below 75 mg/dL, the within-run and between standard deviation (SD) will be computed; for levels with targets great than or equal to 75 mg/dL, the coefficient of variation (CV) will be computed, using the average over all runs.

Scatterplots of control result against targets, together with regression lines, for each instrument will be constructed. The Differences from target will be plotted against the target values for each instrument.

#### 13. Meter Control Solution Results

Each meter unit used in the study will have control solution tests performed. The acceptable range of control solution results is specific to each meter, and the limits are provided by R&D or Quality Assurance. The control solution results must fall within prescribed limits in order for a meter to be used in the study. There are up to 3 attempts allowed to obtain a within-limit result for each meter.

## **Mock Tables and Graphs**

Mock tables and graphs are intended to illustrate the general nature of such tables and graphs that are to be included in the study report. As such, they are facsimiles; actual tables and graphs may vary from the mock versions. For example, studies may have more than one site. The actual tables indicating results are computed by site would have results for each site included in the study.

Section 3 – Proportions: Applies to Sections 3.1-3.3, 3.5, 3.7

Table 3.1. Proportion -15 mg/dL  $\leq$  D  $\leq$  +15 mg/dL (LabBG < 100 mg/dL) or -15%  $\leq$  RD  $\leq$  +15% (LabBG  $\geq$  100 mg/dL)

| Level | Count | Percent | Lower CI | Upper CI | 1-Alpha |
|-------|-------|---------|----------|----------|---------|
| ln | 317 | 97.84% | 95.61% | 98.95% | 0.95 |
| Out | 7 | 2.16% | 1.05% | 4.39% | 0.95 |
| Total | 324 | | | | |

Section 3 – Descriptive Statistics for D, RD

Table 3.2. Descriptive Statistics for D and RD

| Level mg/dL | Variable | N | Mean | Std Dev | Min | Max | Median |
|--------------|-----------|-----|------|---------|--------|-------|--------|
| LT 100 | D (mg/dL) | 74 | 2.19 | 4.470 | -12.40 | 15.20 | 2.75 |
| GE 100 | RD (%) | 297 | 3.17 | 4.945 | -28.09 | 25.36 | 3.23 |
| Level mmol/L | Variable | Ν | Mean | Std Dev | Min | Max | Median |
| LT 5.55 | D (mg/dL) | 74 | 0.12 | 0.25 | -0.69 | 0.84 | 0.15 |
| GE 5.55 | RD (%) | 297 | 3.17 | 4.945 | -28.09 | 25.36 | 3.23 |

# Section 4 – Regression Plot

**Table 4.1 Regression Statistics** 

| Variable | Term | Estimate | Std Error | LCL | UCL | Adj. R <sup>2</sup> | RMSE | d.f.e. |
|---|---|---|---|---|---|---|---|---|
| Sub.Cap. | Intercept | 1.253 | 0.9989 | -0.712 | 3.218 | 0.9827 | 0.0481 | 322 |
| | YSICAP | 1.024 | 0.0076 | 1.009 | 1.039 | | | 322 |
| AST | Intercept | 0.834 | 1.3671 | -1.856 | 3.524 | 0.9672 | 0.0663 | 323 |
| | YSICAP | 1.008 | 0.0103 | 0.988 | 1.029 | | | 323 |
| Staff Test | Intercept | -0.776 | 0.8393 | -2.427 | 0.875 | 0.9882 | 0.0405 | 322 |
| | YSICAP | 1.044 | 0.0063 | 1.032 | 1.057 | | | 322 |
| Venous | Intercept | 3.035 | 1.6399 | -0.192 | 6.261 | 0.9506 | 0.0819 | 316 |
| | YSIVEN | 0.988 | 0.0127 | 0.963 | 1.013 | | | 316 |
| | Estimate = | = Least Squ | ares Value | | | | | |
| | Std Error = | Standard | Error of Est | timate | | | | |
| | LCL = Low | er Confide | nce Limit | | | | | |
| | UCL = Upp | er Confide | nce Limit | | | | | |
| | Adj. $R^2 = A$ | Adjusted R- | squared | | | | | |
| | RMSE = Ro | ot Mean S | quare Erro | r | | | | |
| | d.f.e. = De | grees of F | reedom fo | r Error | | | | |

Figure 4.1. Regression Plot



Section 4 – Modified Bland-Altman Plot

Figure 4.2. Modified Bland-Altman Plot



Note: D-SCP-O represents differences (D) for points identified as outliers; D-SCP-N are non-outlier points. LL-diff and UL-diff are the ISO 15197:2013, section 8 limits on accuracy.

Section 5 – Consensus (Parkes) Error Grid

Figure 5.1. Parkes Error Grid

# GCA-PRO-2014-002-01 Karajishi Contour(R) - Staff Capillary

**Parkes Error Grid Analysis** 

| Zone | A | В | С | D | Е |
|---|---|---|---|---|---|
| Freq | Freq 326 out of 326 0 out of 32 | | 0 out of 326 | 0 out of 326 | 0 out of 326 |
| %Freq | 100.0% | 0.0% | 0.0% | 0.0% | 0.0% |



# Section 7 – Subject Questionnaires

**Table 7.1. Ease of Use Statements** 

| Statement No. | Ease of Use |
|---|---|
| S1 | I find it easy to do a fingerstick blood test with this meter. |
| S2 | The meter display is easy to see and read. |
| S3<br>S4 | It was easy to understand my test results. |
| S4 | I like the overall meter design. |
| S5 | I find the meter easy to use. |
| S6 | The instructions (User Guide and Quick Reference Guide) were easy to understand. |
| S7 | The instructions clearly explain how to run a test. |
| S8 | The instructions clearly explain what to do if an error message is displayed by the meter. |

**Table 7.2.** Ease of Use Results

Note: columns labeled  $\% \ge$  Neutral and Crit. % will not appear in the table for the FDA report.

| | Strongly | | | | Strongly | Total No. | %≥ | |
|---|---|---|---|---|---|---|---|---|
| | Disagree | Disagree | Neutral | Agree | Agree | <b>A</b> nswered | Neutral | Crit. % |
| S1 | 1 | 3 | 19 | 98 | 251 | 372 | 98.92% | 87.63% |
| S2 | 1 | 0 | 1 | 76 | 294 | 372 | 99.73% | 87.63% |
| S3 | 1 | 0 | 11 | 64 | 296 | 372 | 99.73% | 87.63% |
| S4 | 2 | 2 | 39 | 125 | 204 | 372 | 98.92% | 87.63% |
| S5 | 1 | 2 | 11 | 93 | 265 | 372 | 99.19% | 87.63% |
| S6 | 2 | 2 | 31 | 105 | 232 | 372 | 98.92% | 87.63% |
| S7 | 1 | 3 | 10 | 92 | 266 | 372 | 98.92% | 87.63% |
| S8 | 1 | 0 | 17 | 98 | 256 | 372 | 99.73% | 87.63% |

**Table 7.3. Diabetes Management Statements** 

| Table 7.5. Dia | betes Management Statements |
|---|---|
| | Diabetes Mgt. Survey (PWDs Only) |
| Statement No. | Accuracy is important to help with: |
| S1 | 1a) My ability to talk with my Health Care Professional |
| S2 | 1b) My satisfaction with my self-monitoring of diabetes. |
| S3 | 1c) My ability to manage my diabetes. |
| S4 | 1d) Preventing low blood sugars. |
| S5 | 1e) Understanding how food or exercise affects low blood sugars. |
| S6 | 1f) Using my results to gain better control of my diabetes. |
| S7 | 1g) Achieving greater peace of mind. |
| S8 | 2. I prefer the meter that I just used to my regular meter |
| | I use my current meter because: |
| S9 | 3a) My care provider gave it to me |
| S10 | 3b) My insurance company covers the strips |
| S11 | 3c) I think it is the most accurate meter |

**Table 7.4. Diabetes Management Results** 

| | | | S | COR | Ε | | |
|-------------|----|----|----|-----|----|-----|--------|
| Statement | 0 | 1 | 2 | 3 | 4 | 5 | Total* |
| Question 1 | 3 | 0 | 0 | 12 | 54 | 263 | 329 |
| Question 2 | 2 | 0 | 1 | 4 | 64 | 261 | 330 |
| Question 3 | 1 | 0 | 2 | 6 | 53 | 270 | 331 |
| Question 4 | တ | 0 | 1 | 9 | 63 | 250 | 323 |
| Question 5 | 2 | 0 | 1 | 8 | 58 | 263 | 330 |
| Question 6 | 0 | 0 | 2 | 1 | 48 | 281 | 332 |
| Question 7 | 2 | 1 | 2 | 10 | 67 | 250 | 330 |
| Question 8 | 16 | 12 | 13 | 95 | 75 | 121 | 316 |
| Question 9 | 40 | 22 | 21 | 21 | 67 | 161 | 292 |
| Question 10 | 26 | 28 | 16 | 18 | 55 | 189 | 306 |
| Question 11 | 24 | 16 | 33 | 135 | 76 | 48 | 308 |

<sup>\*</sup>Total number of subjects who responded

Section 8all of these tables below are needed for ALL and only PWD

**Table 8.1. Ethnicity** 

| Ethnicity | Count | Percent |
|------------------------|-------|---------|
| Hispanic or Latino | 47 | 12.63% |
| Not Hispanic or Latino | 320 | 86.02% |
| Not Reported | 5 | 1.34% |
| Total | 372 | 100.00% |

Table 8.2. Race

| Race | Count | Percent |
|---------------------------|-------|---------|
| White | 305 | 81.99% |
| Black | 32 | 8.60% |
| Asian | 23 | 6.18% |
| Native American | 7 | 1.88% |
| Hawaiian/Pacific Islander | 4 | 1.08% |
| Not Reported | 7 | 1.88% |

Table 8.3. Languages Spoken

| Laguage Spoken | Count | Percent |
|----------------|-------|---------|
| English | 363 | 97.58% |
| Spanish | 10 | 2.69% |
| BUNGABA | 1 | 0.27% |
| HINDI, PUNJABI | 1 | 0.27% |
| KANNADA | 1 | 0.27% |
| TAGALOG | 2 | 0.54% |
| URDU | 2 | 0.54% |
| VIETNAMESE | 1 | 0.27% |

**Table 8.4. Education** 

| Education | Count | Percent |
|------------------------------------|-------|---------|
| Bachelors degree or more | 110 | 29.57% |
| High school graduate or equivalent | 66 | 17.74% |
| Less than high school | 7 | 1.88% |
| Not reported | 2 | 0.54% |
| Some college or Associate degree | 187 | 50.27% |
| Total | 372 | 100.00% |

Table 8.5. Occupation

| Occupation | Count | Percent |
|-------------------|-------|---------|
| Administrative | 109 | 29.30% |
| Manufacturing | 43 | 11.56% |
| Professional | 113 | 30.38% |
| Sales/Services | 122 | 32.80% |
| Student | 74 | 19.89% |
| Retired | 96 | 25.81% |
| Health Care Field | 53 | 14.25% |
| Work at home | 51 | 13.71% |
| Other | 42 | 11.29% |
| Not reported | 2 | 0.54% |

Table 8.6. Gender

| Gender | Count | Percent |
|--------|-------|---------|
| Female | 201 | 54.03% |
| Male | 171 | 45.97% |
| Total | 372 | 100.00% |

**Table 8.7. Age Statistics** 

| N | Mean | SD | Median | Min | Max | # < 65 | % < 65 |
|-----|------|-------|--------|-----|-----|--------|--------|
| 376 | 52.1 | 15.60 | 55 | 18 | 81 | 295 | 78.46% |

Table 8.8. Diabetes Type

| Table 6.6. Diabetes Type | | |
|-------------------------------|-------|---------|
| Туре | Count | Percent |
| Do not have diabetes | 43 | 11.56% |
| Don't know (Type 1 or Type 2) | 3 | 0.81% |
| Type 1 | 121 | 32.53% |
| Type 2 | 205 | 55.11% |
| Total | 372 | 100.00% |

Table 8.9. Diabetes History (PWD Subjects Only)

| Variable | Level | Count | Percent |
|-------------|--------------------------------------|-------|---------|
| Time | 1 to 3 months | 6 | 1.82% |
| Since | 4 to 6 months | 1 | 0.30% |
| Diagnosis | 7 to 12 months | 3 | 0.91% |
| | 13 months to 2 years | 22 | 6.69% |
| | 3 to 5 years | 25 | 7.60% |
| | 6 to 10 years | 58 | 17.63% |
| | More than 10 years | 214 | 65.05% |
| | Total | 329 | 100.00% |
| Testing | 1 time per day | 54 | 16.41% |
| Frequency | 2 times per day | 63 | 19.15% |
| | 3 times per day | 49 | 14.89% |
| | 4 times per day | 35 | 10.64% |
| | I don't test my blood glucose | 11 | 3.34% |
| | Less than 1 time per day | 39 | 11.85% |
| | More than 4 times per day | 78 | 23.71% |
| | Total | 329 | 100.00% |
| Recommended | 1 time per day | 57 | 17.33% |
| Testing | 2 times per day | 55 | 16.72% |
| Frequency | 3 times per day | 61 | 18.54% |
| | 4 times per day | 52 | 15.81% |
| | Less than 1 time per day | 10 | 3.04% |
| | More than 4 times per day | 81 | 24.62% |
| | My HCP does not recommend BG testing | 13 | 3.95% |
| | Total | 329 | 100.00% |
| Insulin | Insulin pump | 75 | 35.21% |
| Use | One or two injections per day | 57 | 26.76% |
| Frequency | Three or more injections per day | 81 | 38.03% |
| | Total | 213 | 100.00% |

Table 8.9. Diabetes History Continued (PWD Subjects Only)

| Variable | Level | Count | Percent |
|-------------|----------------------------------------------|-------|---------|
| HbA1c | 6.0 % or lower | 23 | 6.99% |
| | 6.1 to 6.5 % | 37 | 11.25% |
| | 6.6 to 7.0 % | 48 | 14.59% |
| | 7.1 to 7.5 % | 63 | 19.15% |
| | 7.6 to 8.0 % | 32 | 9.73% |
| | 8.1 to 8.5 % | 25 | 7.60% |
| | 8.6 to 9.0 % | 8 | 2.43% |
| | 9.1 to 9.5 % | 17 | 5.17% |
| | 9.6 to 10.0 % | 7 | 2.13% |
| | 10.1 to 10.5 % | 2 | 0.61% |
| | Greater than 10.5 % | 14 | 4.26% |
| | I don't know | 52 | 15.81% |
| | I have never gotten an A1C test | 1 | 0.30% |
| | Total | 329 | 100.00% |
| Type of HCP | Diabetologist | 1 | 0.30% |
| | Endocrinologist | 149 | 45.29% |
| | General/ Family practitioner | 159 | 48.33% |
| | Internist | 12 | 3.65% |
| | Other | 8 | |
| | Total | 329 | 100.00% |
| Other HCP | ARNP | 1 | 12.50% |
| | COMMUNITY CLINIC | 1 | 12.50% |
| | D.0 | 1 | 12.50% |
| | INTERNAL MEDICINE | 1 | 12.50% |
| | NURSE PRACTITIONER | 2 | 25.00% |
| | P.A. | 1 | 12.50% |
| | RN | 1 | 12.50% |
| | Total | 8 | 100.00% |
| Use | I do not know what DMS is | 12 | 3.65% |
| Data Mgt. | No | 259 | 78.72% |
| Software | No (do NOT use at home) | 29 | |
| | Yes | 29 | 8.82% |
| | Total | 329 | 100.00% |
| DM Software | Daily | 2 | 6.90% |
| Frequency | Less than monthly | 4 | 13.79% |
| of Use | Monthly | 6 | |
| | Only in preparation for Doctor's appointment | 14 | 48.28% |
| | Weekly | 3 | |
| | Total | 29 | 100.00% |

Table 8.9. Diabetes History Continued (PWD Subjects Only)

| Adjust Therapy | No | 123 | 37.39% |
|----------------|-------|-----|---------|
| based on | Yes | 206 | 62.61% |
| BG Results? | Total | 329 | 100.00% |
| Manage | No | 116 | 35.26% |
| Diabetes with | Yes | 213 | 64.74% |
| Insulin? | Total | 329 | 100.00% |

Table 8.10. Subjects Taking Pre-Defined List of Medications

| Subject take any | | |
|------------------|-------|---------|
| Drugs Listed? | Count | Percent |
| No | 17 | 4.57% |
| Yes | 355 | 95.43% |
| Total | 372 | 100.00% |

Table 8.11. Numbers and Percents of Subjects Taking Pre-Defined Medications

| <b>Abbreviation</b> | Drug Name | Count | Percent |
|---------------------|---------------------------|-------|---------|
| AMARYL | Amaryl / Glimepiride | 7 | 1.88% |
| ASPIRIN | Aspirin | 163 | 43.82% |
| COFFEE | Coffee / Caffeine | 291 | 78.23% |
| EPHEDRIN | Ephedrine/ (Sudafed) | 19 | 5.11% |
| GLUCOPHA | Glucophage / Metformin | 159 | 42.74% |
| GLUCOTRO | Glucotrol / Glipizide | 19 | 5.11% |
| MICRONAS | Micronase /Glyburide | 7 | 1.88% |
| MOTRIN | Motrin/Ibuprofen | 139 | 37.37% |
| PIOGLITA | Pioglitazone / Actos | 4 | 1.08% |
| TETRACYC | Tetracycline | 1 | 0.27% |
| TYLENOL | Tylenol / Acetaminophen | 98 | 26.34% |
| VITAMINC | Vitamin C / Ascorbic Acid | 93 | 25.00% |
| None | None | 17 | 4.57% |

Table 8.12. No. PWD Subjects with Pre-Defined Conditions

| | No. PWD | No. | |
|------------------------|-------------|-----|--------|
| Condition: | w/Condition | PWD | % PWD |
| Have any of following? | 209 | 329 | 63.53% |
| Parkinson's | 0 | 329 | 0.00% |
| Liver Disease | 2 | 329 | 0.61% |
| Kidney Disease | 14 | 329 | 4.26% |
| Hyperlipidemia | 146 | 329 | 44.38% |
| Gout | 16 | 329 | 4.86% |
| Hypertension | 154 | 329 | 46.81% |
| Cardiac Disease | 19 | 329 | 5.78% |

Table 8.13. No. Non-PWD Subjects with Pre-Defined Conditions

| | No. Non-PWD | No. | |
|------------------------|-------------|---------|-----------|
| Condition: | w/Condition | Non-PWD | % Non-PWD |
| Have any of following? | 8 | 43 | 18.60% |
| Parkinson's | 0 | 43 | 0.00% |
| Liver Disease | 1 | 43 | 2.33% |
| Kidney Disease | 0 | 43 | 0.00% |
| Hyperlipidemia | 6 | 43 | 13.95% |
| Gout | 0 | 43 | 0.00% |
| Hypertension | 2 | 43 | 4.65% |
| Cardiac Disease | 0 | 43 | 0.00% |

Table 8.14. No. All Types of Subjects with Pre-Defined Conditions

| | No. ANY | No. | |
|------------------------|-------------|-------|---------|
| Condition: | w/Condition | Total | % Total |
| Have any of following? | 217 | 372 | 58.33% |
| Parkinson's | 0 | 372 | 0.00% |
| Liver Disease | 3 | 372 | 0.81% |
| Kidney Disease | 14 | 372 | 3.76% |
| Hyperlipidemia | 152 | 372 | 40.86% |
| Gout | 16 | 372 | 4.30% |
| Hypertension | 156 | 372 | 41.94% |
| Cardiac Disease | 19 | 372 | 5.11% |

Section 9 – Other Tables – 9.1 and 9.3

Table 9.1. LabBG and HCT Descriptive Statistics

| Variable | Population | Site | N | Mean | SD | Median | Min | Max | < 80 | > 250 |
|---|---|---|---|---|---|---|---|---|---|---|
| YSI CAP | PWD | 1 | 163 | 152.80 | 65.214 | 139.50 | 44.95 | 455.50 | 11 | 14 |
| YSI CAP | PWD | 2 | 169 | 155.92 | 75.237 | 135.50 | 32.25 | 458.00 | 11 | 17 |
| YSI CAP | PWD | Both | 332 | 154.39 | 70.405 | 136.00 | 32.25 | 458.00 | 22 | 31 |
| YSI CAP | ALL | 1 | 184 | 146.23 | 64.330 | 126.75 | 44.95 | 455.50 | 11 | 14 |
| YSI CAP | ALL | 2 | 191 | 148.71 | 73.586 | 127.50 | 32.25 | 458.00 | 11 | 17 |
| YSI CAP | ALL | Both | 375 | 147.49 | 69.119 | 127.50 | 32.25 | 458.00 | 22 | 31 |
| Hematocrit | PWD | 1 | 163 | 43.09 | 4.036 | 43 | 34 | 59 | | |
| Hematocrit | PWD | 2 | 169 | 43.44 | 3.767 | 44 | 33 | 52 | | |
| Hematocrit | PWD | Both | 332 | 43.27 | 3.899 | 43 | 33 | 59 | | |
| Hematocrit | ALL | 1 | 184 | 43.02 | 3.939 | 43 | 34 | 59 | | |
| Hematocrit | ALL | 2 | 191 | 43.41 | 3.742 | 43 | 33 | 52 | | |
| Hematocrit | ALL | Both | 375 | 43.22 | 3.840 | 43 | 33 | 59 | | |
| YSI VEN | PWD | 1 | 162 | 149.18 | 65.075 | 136.50 | 47.30 | 455.00 | 15 | 12 |
| YSI VEN | PWD | 2 | 168 | 152.58 | 75.251 | 131.25 | 30.25 | 461.00 | 16 | 16 |
| YSI VEN | PWD | Both | 330 | 150.91 | 70.353 | 133.50 | 30.25 | 461.00 | 31 | 28 |

Note: HCT = hematocrit; YSI = capillary YSI LabBG; YSI-VEN = venous YSI LabBG

Section 9 – Temperature (Temp) and Relative Humidity (RH)

**Table 9.2. Temperature and Relative Humidity** 

| Site | Variable | Ν | Mean | SD | Median | Min | Max |
|------|-----------------------|----|-------|-------|--------|------|------|
| 1 | Temperature (°F) | 28 | 70.42 | 0.581 | 70.4 | 68.5 | 71.8 |
| 2 | Temperature (°F) | 44 | 72.08 | 0.965 | 72.3 | 70.0 | 74.7 |
| 1 | Relative Humidity (%) | 28 | 36.89 | 5.370 | 39.0 | 24.0 | 44.0 |
| 2 | Relative Humidity (%) | 44 | 37.34 | 4.467 | 37.0 | 27.0 | 47.0 |
| Both | Temperature (°F) | 72 | 71.43 | 1.164 | 71.5 | 68.5 | 74.7 |
| Both | Relative Humidity (%) | 72 | 37.17 | 4.806 | 38.0 | 24.0 | 47.0 |

# Section 11 – Evaluability

**Table 11.1. Numbers of Non-Evaluables** 

| RESULT TYPE | Total No. Subjects | Non-eval | Missing Meter BG | No HCT | Usable N |
|---|---|---|---|---|---|
| SUBJECT RESULT | 372 | 1 | 5 | 1 | 365 |
| STUDY STAFF RESULT | 372 | 1 | 1 | 1 | 369 |
| Non-PWD-SUB | 43 | 0 | 2 | 0 | 41 |
| Non-PWD-STAFF | 43 | 0 | 0 | 0 | 43 |
| Total PWDs | 329 | | | | |
| PWDs used for ISO-SUB CAP | | | | | 324 |
| PWDs used for ISO-STAFF CAP | | | | | 326 |
| VENOUS | 329 | 0 | 10 | 1 | 318 |
| Note: 3006 had missing venous BG | CT | | | | |

# Section 12 – Laboratory Instrument Quality Control

**Table 12.1. Accuracy Statistics** 

| | | | | | D = YSI - T | ) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site | YSINUM | LEVEL | Target | N | Mean(D) | Std Dev(D) | Median(D) | Min(D) | Max(D) |
| 1 | 10 | 2 | 50.0 | 38 | -0.44 | 0.606 | -0.40 | -1.60 | 0.70 |
| 1 | 10 | 3 | 98.5 | 38 | 0.05 | 1.023 | 0.35 | -1.90 | 1.50 |
| 1 | 10 | 4 | 197.3 | 38 | -1.35 | 1.355 | -1.30 | -3.30 | 1.70 |
| 1 | 10 | 5 | 394.5 | 38 | -1.87 | 3.560 | -2.50 | -8.50 | 4.50 |
| 1 | 11 | 2 | 50.0 | 38 | -0.73 | 0.812 | -0.70 | -2.40 | 1.60 |
| 1 | 11 | 3 | 98.5 | 38 | -0.50 | 1.400 | -0.20 | -3.40 | 1.50 |
| 1 | 11 | 4 | 197.3 | 38 | -2.09 | 2.055 | -1.80 | -5.30 | 1.70 |
| 1 | 11 | 5 | 394.5 | 38 | -3.79 | 3.631 | -3.50 | -15.50 | 2.50 |
| 2 | 48 | 2 | 50.0 | 34 | -1.24 | 0.595 | -1.30 | -2.20 | 0.00 |
| 2 | 48 | 3 | 98.5 | 34 | -1.52 | 1.402 | -1.45 | -4.30 | 1.00 |
| 2 | 48 | 4 | 197.3 | 34 | -3.56 | 2.300 | -3.80 | -7.30 | 0.70 |
| 2 | 48 | 5 | 394.5 | 34 | -3.82 | 3.169 | -4.00 | -9.50 | 4.50 |
| 2 | 98 | 2 | 50.0 | 34 | -1.30 | 0.535 | -1.20 | -2.30 | -0.20 |
| 2 | 98 | 3 | 98.5 | 34 | -1.42 | 1.431 | -1.35 | -4.30 | 1.00 |
| 2 | 98 | 4 | 197.3 | 34 | -4.01 | 1.915 | -4.30 | -8.30 | -0.30 |
| 2 | 98 | 5 | 394.5 | 34 | -3.94 | 3.067 | -4.00 | -10.50 | 1.50 |

| | | | | | RD = 100( | YSI - Target)/ | Γarget (%) | | |
|---|---|---|---|---|---|---|---|---|---|
| Site | YSINUM | LEVEL | Target | N | Mean(RD) | Std Dev(RD) | Median(RD) | Min(RD) | Max(RD) |
| 1 | 10 | 2 | 50.0 | 38 | -0.88 | 1.212 | -0.80 | -3.20 | 1.40 |
| 1 | 10 | 3 | 98.5 | 38 | 0.05 | 1.039 | 0.36 | -1.93 | 1.52 |
| 1 | 10 | 4 | 197.3 | 38 | -0.69 | 0.687 | -0.66 | -1.67 | 0.86 |
| 1 | 10 | 5 | 394.5 | 38 | -0.47 | 0.902 | -0.63 | -2.15 | 1.14 |
| 1 | 11 | 2 | 50.0 | 38 | -1.47 | 1.624 | -1.40 | -4.80 | 3.20 |
| 1 | 11 | 3 | 98.5 | 38 | -0.50 | 1.421 | -0.20 | -3.45 | 1.52 |
| 1 | 11 | 4 | 197.3 | 38 | -1.06 | 1.042 | -0.91 | -2.69 | 0.86 |
| 1 | 11 | 5 | 394.5 | 38 | -0.96 | 0.920 | -0.89 | -3.93 | 0.63 |
| 2 | 48 | 2 | 50.0 | 34 | -2.48 | 1.190 | -2.60 | -4.40 | 0.00 |
| 2 | 48 | 3 | 98.5 | 34 | -1.54 | 1.424 | -1.47 | -4.37 | 1.02 |
| 2 | 48 | 4 | 197.3 | 34 | -1.81 | 1.166 | -1.93 | -3.70 | 0.35 |
| 2 | 48 | 5 | 394.5 | 34 | -0.97 | 0.803 | -1.01 | -2.41 | 1.14 |
| 2 | 98 | 2 | 50.0 | 34 | -2.60 | 1.070 | -2.40 | -4.60 | -0.40 |
| 2 | 98 | 3 | 98.5 | 34 | -1.44 | 1.452 | -1.37 | -4.37 | 1.02 |
| 2 | 98 | 4 | 197.3 | 34 | -2.03 | 0.971 | -2.18 | -4.21 | -0.15 |
| 2 | 98 | 5 | 394.5 | 34 | -1.00 | 0.777 | -1.01 | -2.66 | 0.38 |

**Table 12.2. Precision Statistics** 

| LEVEL | YSINUM | Random Effect | Mean | SigEst | CV |
|-------|--------|---------------|--------|--------|-------|
| 2 | 10 | Between | 49.56 | 0.604 | 1.22% |
| 2 | 10 | Within | 49.56 | 0.111 | 0.22% |
| 2 | 10 | Total | 49.56 | 0.614 | 1.24% |
| 3 | 10 | Between | 98.55 | 1.027 | 1.04% |
| 3 | 10 | Within | 98.55 | 0.147 | 0.15% |
| 3 | 10 | Total | 98.55 | 1.037 | 1.05% |
| 4 | 10 | Between | 195.95 | 1.333 | 0.68% |
| 4 | 10 | Within | 195.95 | 0.324 | 0.17% |
| 4 | 10 | Total | 195.95 | 1.372 | 0.70% |
| 5 | 10 | Between | 392.63 | 3.533 | 0.90% |
| 5 | 10 | Within | 392.63 | 0.725 | 0.18% |
| 5 | 10 | Total | 392.63 | 3.607 | 0.92% |
| 2 | 11 | Between | 49.27 | 0.806 | 1.64% |
| 2 | 11 | Within | 49.27 | 0.165 | 0.33% |
| 2 | 11 | Total | 49.27 | 0.823 | 1.67% |
| 3 | 11 | Between | 98.00 | 1.401 | 1.43% |
| 3 | 11 | Within | 98.00 | 0.223 | 0.23% |
| 3 | 11 | Total | 98.00 | 1.419 | 1.45% |
| 4 | 11 | Between | 195.21 | 2.044 | 1.05% |
| 4 | 11 | Within | 195.21 | 0.397 | 0.20% |
| 4 | 11 | Total | 195.21 | 2.083 | 1.07% |
| 5 | 11 | Between | 390.71 | 3.573 | 0.91% |
| 5 | 11 | Within | 390.71 | 0.874 | 0.22% |
| 5 | 11 | Total | 390.71 | 3.678 | 0.94% |

Figure 12.1. Scatterplot with Regression Line





Figure 12.2. Difference from Target Plot (for YSI Control Solution Tests)



Diff = control result - target

**Table 12.3. Regression Statistics** 

| Site | Term | Estimate | Std Error | d.f.e. | LCL | UCL | Adj. R <sup>2</sup> | Sy.x |
|---|---|---|---|---|---|---|---|---|
| 1 | Intercept | -0.212 | 0.1029 | 302 | -0.415 | -0.010 | 0.9996 | 0.0120 |
| 1 | Slope | 0.995 | 0.0012 | 302 | 0.992 | 0.997 | 0.9996 | 0.0120 |
| 2 | Intercept | -0.710 | 0.1057 | 270 | -0.918 | -0.502 | 0.9996 | 0.0117 |
| 2 | Slope | 0.989 | 0.0012 | 270 | 0.987 | 0.992 | 0.9996 | 0.0117 |

Section 13 – Meter Controls

**Table 13.1. Meter Control Results Summary** 

| Site | Lot | Ν | Mean | SD | Median | Min | Max | LL | UL |
|---|---|---|---|---|---|---|---|---|---|
| 1 | BLUE | 20 | 126.6 | 2.19 | 126.0 | 123 | 132 | 110 | 138 |
| 1 | GREEN | 20 | 128.0 | 2.31 | 128.0 | 124 | 131 | 110 | 137 |
| 1 | RED | 20 | 129.0 | 1.79 | 129.0 | 125 | 131 | 109 | 136 |
| 2 | BLUE | 20 | 121.2 | 2.07 | 121.0 | 117 | 125 | 110 | 138 |
| 2 | <b>GREEN</b> | 20 | 123.2 | 1.79 | 122.5 | 121 | 127 | 110 | 137 |
| 2 | RED | 20 | 121.7 | 1.72 | 122.0 | 118 | 125 | 109 | 136 |
| LL = Lower Limit | | | | | | | | | |
| UL = Upper Limit | | | | | | | | | |